CLINICAL TRIAL: NCT01671176
Title: A Clinical Study of the Oticon Medical Ponto 4.5mm Wide Implant
Brief Title: Wide Diameter Bone Anchored Implant Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Wide04262012
Record Dates: First submitted 2012-08-15; First posted 2012-08-23 (Estimated); Results first posted 2018-05-07 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-04

CONDITIONS: Conductive Hearing Loss; Conductive and Sensori-neural Hearing Loss in the Same Ear; Unilateral, Profound Sensori-neural Hearing Loss
Keywords: Wide diameter implant; ISQ; Ponto; Bone anchored implant
MeSH Terms: conditions — Hearing Loss, Conductive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Wide diameter bone anchored implant (Other): Intervention: Implantation of a wide diameter bone anchored auditory implant either 3 or 4 mm in length, into the skull on the side of the ear where intervention is intended in order to restore hearing. In the case of a conductive or mixed hearing loss, that side is chosen. In patients with unilateral, profound sensori-neural hearing loss the implant is implanted on that side but the sound is transmitted to the side with the normal hearing ear via bone conduction stimulation.
  Interventions: Device: Wide diameter bone anchored implant

INTERVENTIONS:
Device: Wide diameter bone anchored implant — 4.5 mm wide diameter bone anchored implant
  Other Names: Oticon Medical Ponto Pro; Oticon Medical Ponto Pro Power; Osstell ISQ

SUMMARY:
To assess implant stability, implant loss, adverse skin reactions, and Quality of Life Benefit following implantation of the Ponto 4.5mm Wide Diameter implant. Secondary: to determine the feasibility of fitting the sound processor 3 weeks after surgical implantation, and to investigate if the type of skin reactions following implantation could be related to the demographic data of subjects and the type of surgical technique used

DETAILED DESCRIPTION:
Bone-anchored hearing systems have been an amplification choice for conductive, mixed, and profound, unilateral, sensorineural hearing loss for over three decades. So far, about 75,000 patients worldwide have received this surgical intervention (bone-anchored hearing system), since its first successful implantation in 1977. In 2009, Oticon Medical, LLC launched its bone-anchored hearing system called Ponto. In just over two years, the Ponto has been successfully implanted in over 3,000 patients by leading otolaryngologists and neurotologists in 18 countries worldwide.

The Ponto implant has previously been available with a 3.75mm diameter and comes in two lengths: 3mm and 4mm. Anew Ponto implant that is 4.5mm wide in diameter is now available in both 3mm and 4mm lengths. This Wide Diameter implant is designed to maximize bone-to-implant contact area and enhance implant stability which can potentially allow loading of the sound processor as early as 3 weeks after surgery. The abutment screw incorporates external threads at the screw head to make it possible to connect a SmartPeg (Osstell, Goteborg, Sweden) for stability measurements. All Ponto implants have the same universal implant-abutment interface. Therefore, they are fully compatible with existing instruments and abutments. Two new countersinks have been developed for the new Ponto Wide Diameter implant. The drill size of the countersink is 3.80mm. It is marked with a "W" to separate them from existing drills. All products are CE-marked and cleared for the US market by the FDA.

Objectives The present study will attempt to show that the Ponto 4.5mm Wide Diameter implant has similar or better outcomes in terms of Quality of Life (QoL) benefit; implant extrusion and revision surgery when compared to the 3.75mm diameter implant. Secondary objectives to be studied will include adverse skin reactions, the feasibility of fitting the sound processor three weeks after surgical implantation, and investigation to see if the type of skin reactions observed following implantation could be related to the demographic data of subjects or the type of surgical technique used.

Study Design This study is a prospective, multicenter study of subjects' demographic and implant data. Subjects will be enrolled at two US sites.

Subject Population Twenty adult subjects 18 years or older will be included in the study from each participating partner site.

ELIGIBILITY:
Inclusion Criteria:

* conductive, mixed or single sided deafness
* 18 years of age or older

Exclusion Criteria:

* younger than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack Wazen, MD, Principal Investigator — Sarasota Ear Institute
Locations (2):
- United States (2):
  - Silverstein Institute, Sarasota, Florida
  - Michigan Ear Institute, Farmington Hills, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wazen JJ, Babu S, Daugherty J, Metrailer A. Three-week loading of the 4.5mm wide titanium implant in bone anchored hearing systems. Am J Otolaryngol. 2016 Mar-Apr;37(2):132-5. doi: 10.1016/j.amjoto.2015.08.005. Epub 2015 Aug 18. PMID 26954868

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Wide Diameter Bone Anchored Implant
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Wide Diameter Bone Anchored Implant
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.83 (16.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 30
Smoking status [Number; unit: participants]
  yes | 1
  no | 29
Diabetes [Number; unit: participants]
  yes | 3
  no | 27
Abutment length [Number; unit: participants]
  6 mm | 20
  9 mm | 7
  12 mm | 3
Weight [Mean (Standard Deviation); unit: kilogram] | 76.72 (19.61)
BMI [Mean (Standard Deviation); unit: kilogram/M^2] | 28.56 (7.09)
Height [Mean (Standard Deviation); unit: centimeters] | 163.79 (8.89)

OUTCOME MEASURES:

1. Primary Outcome: Holger's Scale
Description: Holger's Scale is a 5 point that ranges from 0 - 4 scale that assesses skin reactions at the implant site where 0 means no reaction and 4 means excessive granulation, skin overgrowth, or scar formation requiring revision surgery
Time Frame: 1 week, 3 weeks, 6 weeks, 3 months, 6 months and 12 months
Measure: Number; unit: participants
Arm/Group | Wide Diameter Bone Anchored Implant
Number analyzed (Participants) | 30
participants
  Holger score 0 at 1 week | 29
  Holger score of 1 at one week | 0
  Holger score of 2 at one week | 1
  Holger score of 0 at 3 weeks | 29
  Holger score of 1 at 3 weeks | 1
  Holger score of 2 at 3 weeks | 0
  Holger score of 0 at 6 weeks | 28
  Holger score of 1 at 6 weeks | 2
  Holger score of 2 at 6 weeks | 0
  Holger score of 0 at 3 months | 29
  Holger score of 1 at 3 months | 1
  Holger score of 2 at 3 months | 0
  Holger score of 0 at 6 months | 30
  Holger score of 1 at 6 months | 0
  Holger score of 2 at 6 months | 0
  Holger score of 0 at 12 months | 29
  olger score of 1 at 12 months 1 | 1
  Holger score of 2 at 12 months | 0

2. Primary Outcome: Implant Stability as Measured by the Osstell Implant Stability Quotient in the Vertical and Horizontal Plane
Description: Presently, the recommendations to load the sound processor on a bone anchored implant is 3 months (for adults). Using outcome measures, i.e., OSSTELL ISQ ranges from 0 -100 where 0 is least stable and 100 being the most stable.
Time Frame: At surgery, 1 week, 3 weeks, 6 weeks, 12 weeks, 6 months and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wide Diameter Bone Anchored Implant
Number analyzed (Participants) | 30
units on a scale
  ISQ vertical at surgery | 58.43 (8.01)
  ISQ horizontal at surgery | 58.58 (7.42)
  ISQ vertical at one week | 59.70 (7.03)
  ISQ horizontal at one week | 59.77 (7.88)
  ISQ vertical at 3 weeks | 60.53 (7.14)
  ISQ horizontal at 3 weeks | 60.30 (7.78)
  ISQ vertical at 6 weeks | 61.28 (5.81)
  ISQ horizontal at 6 weeks | 61.02 (6.56)
  ISQ vertical at 12 weeks | 61.97 (5.91)
  ISQ horizontal at 12 weeks | 62.00 (6.07)
  ISQ vertical at 6 month | 63.62 (5.26)
  ISQ horizontal at 6 months | 63.27 (5.48)
  ISQ vertical at 12 months | 63.73 (5.31)
  ISQ horizontal at 12 months | 63.62 (5.26)

ADVERSE EVENTS:
Arm/Group | Wide Diameter Bone Anchored Implant
Serious Adverse Events (participants affected / at risk) | 1/30
Other Adverse Events (participants affected / at risk) | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Wide Diameter Bone Anchored Implant (N=30)
Skin revision (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No